CLINICAL TRIAL: NCT05357534
Title: Perception of Blood Sugar Variations During Physical Activity in Healthy Subjects and Type 1 Diabetes Patients
Acronym: GLYSPORT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-RIPH_002_GLYSPORT
Record Dates: First submitted 2022-03-21; First posted 2022-05-03 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; blood sugar variations; physical activity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Type 1 diabetes" group (Experimental): "type 1 diabetes" group: patients with type 1 diabetes
  Interventions: Other: Physical activity
- "healthy" group (Active Comparator): "healthy" group : subjects without type 1 diabetes
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — Physical activity: 10 km run on a treadmill

SUMMARY:
Type 1 diabetes is an autoimmune disease with absence of insulin secretion. Blood sugar is a physiological variable that reflets for blood glucose concentration. Blood sugar level fluctuates, especially during physical activity.

Sports activity would increase insulin sensitivity, improve lifestyle and, by extension, promote glycemic balance. However, glycemic balance will be disturbed by physical activity with higher risk of hypoglycemia and hyperglycemia.

Moreover, hypoglycemia and hyperglycemia will impact body functions. Perceptions of blood sugar variations during physical exercise and their influences on sports performance have not been studied, whether in type 1 diabetes patients or healthy subjects.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the perception of blood sugar variations in healthy subjects and type 1 diabetes patients during physical activity

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetics diagnosed more than 3 years ago and controlled (an HbA1c of less than 8%) for "type 1 diabetes" group
* without diabetes for "healkthy" group
* Male
* Aged 18 to 65
* Body Mass Index less than 30 kg/m2
* regular running (at least 30 minutes per week and at least one 10-km run per year for the previous 2 years)
* Agreeing to participate in the study

Exclusion Criteria:

* Physical injury
* beta blockers treatment

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
blood sugar | Day 0
  Blood sugar evaluated in g/L via continuous blood glucose measurement
Feeling lucidity | Day 0
  Lucidity, which is a symptom of hyperglycaemia and hypoglycaemia, assessed by visual analog scale (between "not at all lucid" to "completely lucid"
Feeling fatigue | Day 0
  hydratation, which is a symptom of hyperglycaemia and hypoglycaemia, assessed by visual analog scale (between "no feeling of dehydration" to "dehydrated"
feeling hungry | Day 0
  hungry, which is a symptom of hyperglycaemia and hypoglycaemia, assessed by visual analog scale (between "no feeling of hunger" to "hungry"
average speed per kilometer Sports performance | Day 0
  Sports performance evaluated by average speed per kilometer of the 10 km run on a treadmill
total running time | Day 0
  Sports performance evaluated by total running time of the 10 km run on a treadmill
average running speed | Day 0
  Sports performance evaluated by average running speed of the 10 km run on a treadmill

IPD SHARING:
Plan to Share IPD: No